CLINICAL TRIAL: NCT00900900
Title: The Effects of One-Time Pregnenolone, DHEA, Or Placebo Administration On Withdrawal Symptoms, Mood, Craving And Cigarette Evaluation Ratings In Male Smokers
Brief Title: The Effects of One-Time Pregnenolone, Dehydroepiandrosterone (DHEA), or Placebo Administration On Withdrawal Symptoms, Mood, Craving And Cigarette Evaluation Ratings In Male Smokers
Acronym: DHEA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jed E. Rose (Other)
Responsible Party: Sponsor-Investigator, Jed E. Rose, Professor Department of Psychiatry and Behavorial Sciences, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00008225
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Substance Withdrawal Syndrome
Keywords: Cigarette Smokers; DHEA; dehydroepiandrosterone; pregnenolone; Nicotine withdrawal symptoms
MeSH Terms: conditions — Substance Withdrawal Syndrome | interventions — Dehydroepiandrosterone; Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dehydroepiandrosterone (DHEA) (Experimental)
  Interventions: Dietary Supplement: dehydroepiandrosterone (DHEA)
- Pregnenolone (Experimental)
  Interventions: Dietary Supplement: pregnenolone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: dehydroepiandrosterone (DHEA) — one-time 400mg oral dose of DHEA
  Arms: Dehydroepiandrosterone (DHEA)
Dietary Supplement: pregnenolone — one-time 400mg oral dose of pregnenolone
  Arms: Pregnenolone
Drug: Placebo — one-time dose oral dose
  Arms: Placebo

SUMMARY:
This study will evaluate the potential therapeutic value of two neurosteroid treatments (DHEA and pregnenolone) in the treatment of tobacco withdrawal symptoms. This will include assessing whether these agents relieve craving for cigarettes elicited by exposure to a mildly stressful cognitive task. Pregnenolone (400 mg orally), DHEA (400 mg orally) and placebo will be administered one at each of the three sessions in a randomized order.

ELIGIBILITY:
Inclusion Criteria:

1. male;
2. 18-65 years old;
3. smoked an average of at least 10 cigarettes per day for three cumulative or continuous years of a brand that delivers (by Federal Trade Commission rated yields) at least 0.5 mg nicotine;
4. afternoon expired carbon monoxide reading of at least 10 ppm;
5. in general good health, based on physical examination, EKG serum chemistries, CBC and urinalysis.

Exclusion Criteria:

1. Participants must not have uncontrolled hypertension (systolic >140 mm Hg, diastolic >95 mm Hg)
2. hypotension (systolic <90 mm Hg, diastolic <60 mm Hg);
3. coronary heart disease;
4. heart attack;
5. cardiac rhythm disorder (irregular heart rhythm);
6. chest pains (unless history, exam, and EKG clearly indicate a non-cardiac source);
7. cardiac (heart) disorder (including but not limited to valvular heart disease, heart murmur, heart failure);
8. liver or kidney disorder (except kidney stones, gallstones);
9. gastrointestinal problems or disease other than gastroesophageal reflux,
10. heartburn, or irritable bowel syndrome;
11. ulcers within the past 6 months;
12. lung disorder (including but not limited to COPD, emphysema, and asthma);
13. brain abnormality (including but not limited to, stroke, brain tumor, seizure disorder);
14. history of fainting;
15. problems giving blood samples;
16. diabetes;
17. current cancer or treatment for cancer in the past 6 months (except basal or squamous cell skin cancer);
18. other major medical condition;
19. major depression, panic disorder, anxiety, bipolar disorder, schizophrenia, risk of suicide, or substance dependence other than nicotine dependence;
20. subjects who endorse suicidal ideation on the MINI abridged;
21. alcohol or drugs abuse;
22. reported use of illicit drugs within the past 30 days, or if the drug screen is positive;
23. reported use of smokeless tobacco (chewing tobacco, snuff), cigars, pipes, or nicotine replacement therapy; testosterone replacement therapy, DHEA or Pregnenolone; experimental (investigational) drugs; psychiatric medications (including antidepressants, anti-anxiety agents. anti-psychotics), sleep aids, medications that increase DHEA and/or DHEA-S concentrations (including, but not limited to: diltiazem, benfluorex, amlodipine, alprazolam, danazol, metformin, nitrendipine and retinol), or any other medications that are known to affect smoking (e.g. clonidine, muscle relaxants, opiate pain medications) within the past 2 weeks.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The administration of DHEA or pregnenolone will reduce smoking withdrawal symptoms. | 6 months

SECONDARY OUTCOMES:
The administration of DHEA or pregnenolone will reduce the subjective rewarding effects of nicotine inhaled in cigarette smoke. | 6 months
The administration of DHEA or pregnenolone will reduce stress-induced changes in mood and craving for cigarettes. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jed E Rose, Ph.D., Principal Investigator — Duke University; Christine Marx, M.D., Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke Center for Nicotine & Smoking Cessation Research, Durham, North Carolina
  - Duke Center for Nicotine & Smoking Cessation Research, Raleigh, North Carolina